CLINICAL TRIAL: NCT05191602
Title: A Prospective and Analytical Study on the Detection of Early Anastomotic Leakage With Abdominal Drainage Fluid After Colorectal Cancer Surgery
Brief Title: The Relationship Between Drainage Fluid and Anastomotic Leakage After Colorectal Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Li Chuan, Secretary of General Surgery, Southwest Hospital, China
Other Study IDs: ADFofCRS
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Anastomotic Leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: drainge fluid — including bilirubin

SUMMARY:
A prospective and analytical study on the detection of early anastomotic leakage by abdominal drainage fluid after colorectal cancer surgery. pay attention to indicators including bilirubin

ELIGIBILITY:
Inclusion Criteria:

1) Preoperative pathologically confirmed colorectal adenocarcinoma; 2) Patients undergoing minimally invasive (robot or laparoscopic) tumor resection + bowel anastomosis; 3) Age: 18 to 80 years old; 4) Preoperative TNM staging (whole abdomen) Enhanced CT or MRI, laparoscopic exploration): cT1-3bN0-2M0; 5) Preoperative ASA score: ≤Ⅲ; 6) No history of malignant tumors and no other malignant tumors by preoperative examination; 7) Not accepted before surgery Deterministic treatment, such as radiotherapy, chemotherapy or immunotherapy; 8) No pre-existing ascites was found before and during the operation; 9) Informed consent signed by the patient or his agent

Performance status (ECOG) 0~1

Exclusion Criteria:

1) Patients with obstructive jaundice or other congenital disorders of bile acid synthesis and metabolism; 2) Severe abdominal cavity infection and other infections; 3) A large amount of abdominal effusion was found before and during the operation; 4) Tumor was confirmed during the operation For T4b or intraoperative detection of other tumors, joint resection or distant metastasis is required; 5) Intraoperative conversion to laparotomy; 6) Intraoperative change of surgical method to perform Miles or Hartmann surgery; 7) Intraoperative and postoperative abdominal cavity Hyperthermic perfusion chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
leakage | 10days

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Center of PLA, Chongqing, China